CLINICAL TRIAL: NCT00387283
Title: Pharmacokinetic Study of AVI-4020 in Cerebral Spinal Fluid Among Healthy Adult Males Following Intravenous Administration
Brief Title: Pharmacokinetic Study in Cerebral Spinal Fluid After a Single Dose of AVI-4020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI-4020-21b
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: West Nile Virus
Keywords: WNV; West Nile virus; WNV meningoencephalitis

INTERVENTIONS:
Drug: AVI-4020 Injection

SUMMARY:
During a clinical study of people with severe West Nile virus infections, it was determined that the drug AVI-4020 crossed the blood-brain barrier. This study will assess the amount of drug that goes across the blood-brain barrier and the drug levels measured in both the blood and urine.

The objective of this study is to find out how much and how fast this drug crosses this barrier.

DETAILED DESCRIPTION:
AVI-4020 was designed to interfere with West Nile virus translation, and has been shown to cross the blood-brain barrier in both normal and inflamed meninges in a clinical study in patients with severe West Nile virus disease.

At issue, is whether this observation is limited to AVI-4020 PMO drug, or is observed with other PMO drugs. This study is one of three to assess the specific ability of PMO drugs to cross the blood-brain barrier, using similar dosing, and PK assessment time points. In order to rigorously assess the pharmacokinetics, this study is being performed in healthy volunteers at a single point in time.

The ability of other PMO drugs to cross the blood-brain barrier will set the stage for future studies that exploit this product characteristic.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 18 years to 64 years of age;
* Good general health (as evidenced by no chronic conditions, normal physical exam, vital signs within normal limits; laboratory evaluations within normal range)
* Signed and dated written informed consent form; and
* Willing to participate in all study activities and all requirements, including effective contraception (viz., a double-barrier method) during the 7-day study surveillance period.

Exclusion Criteria:

* Hematology, serum chemistry (exclusive of electrolytes), and urinalysis laboratory test values >2 times upper limits of normal or anemia (hemoglobulin <11 g/dL), leukopenia (total white blood count <3,000/µL or total neutrophils <1,500/ µL) or thrombocytopenia (platelets <100,000/µL). Electrolytes and coagulation values exceeding normal ranges are to be excluded.
* Body Mass Index (BMI) >35.
* Calculated creatinine clearance (by the Cockroft and Gault Formula) <70 mL/min, based on age and gender.
* Positive HIV-1 or HIV-2 serology.
* Positive HCV serology and/or positive plasma HCV-RNA status.
* Positive Hepatitis B status.
* Solid or hematopoetic organ transplant recipient.
* Active illness or recent illness within 30 days of the first dose of study drug.
* History of any of the following: brain injury, neoplasm, chronic or migraine headaches, cancer, meningitis or hydrocephalus.
* Usage of any prescribed, over-the-counter or illicit drug(s) within 30 days of study drug administration. Use of herbal remedies and/or supplements at the discretion of the Investigator.
* Unwilling to practice effective contraception during the study period.
* Participation in any clinical interventional trial within the previous 6 months.
* Positive drug urine screen.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14
Dates: Start 2006-10; Primary Completion 2006-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine if the study drug penetrates the blood brain barrier following a single dose of AVI-4020, and if it does, the associated CSF, plasma and urine pharmacokinetics

SECONDARY OUTCOMES:
Safety, Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Shaw, M.D., Principal Investigator — NW Kinetics
Locations (1):
- NW Kinetics, Tacoma, Washington, United States